CLINICAL TRIAL: NCT03963154
Title: STREAM: A Phase 1/2, Open-label, Safety, Tolerability and Preliminary Efficacy Study of Implantation Into One Eye of hESC-derived RPE in Patients With Retinitis Pigmentosa Due to Monogenic Mutation
Brief Title: Interventional Study of Implantation of hESC-derived RPE in Patients With RP Due to Monogenic Mutation
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre d'Etude des Cellules Souches (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STREAM
Record Dates: First submitted 2019-05-22; First posted 2019-05-24 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Retinitis Pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Intervention Model Description: Open-label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implantation of a therapeutical patch (Experimental): All the patients will receive a single central subretinal implantation in one eye of a monolayer of Human Embryonic Stem Cells-derived Retinal Pigmented Epithelium (hESC-derived RPE). The implanted eye will be the one with the worst visual acuity.
  Interventions: Biological: Human Embryonic Stem Cell Derived Retinal Pigment Epithelium (RPE)

INTERVENTIONS:
Biological: Human Embryonic Stem Cell Derived Retinal Pigment Epithelium (RPE) — Implantation into one eye of hESC-derived RPE (Human Embryonic Stem Cell Derived Retinal Pigment Epithelium (RPE))

SUMMARY:
Phase I/II open-label, safety, tolerability and preliminary efficacy study of implantation into one eye of hESC-derived RPE (Human Embryonic Stem Cell Derived Retinal Pigment Epithelium (RPE)) in patients with retinitis pigmentosa due to monogenic mutation.

Study non randomized single group assignment consisting in 2 sequential cohorts of patients:

* First cohort of 2 patients with very advanced loss of visual acuity (legally blind)
* Second cohort of 10 patients with less advanced loss of visual acuity:

DETAILED DESCRIPTION:
Monocentric study (Hospital of 15-20 at Paris) of duration of 106 weeks.

At total,12 evaluable patients will be enrolled and assigned in 2 cohorts as described above in brief summary.

Expected follow-up for one patient is about 64 weeks including 8 weeks of screening and baseline period and 56 weeks of follow-up after implantation of hESC-derived RPE.

After 56 weeks of follow-up, patients will be enrolled in a long term follow-up study during 4 additional years.

The primary objective is to assess safety and tolerability of implantation of the Investigational Medecinal Product (ISTEM-01) in patients with retinitis pigmentosa.

Secondary objectives are:

* To evaluate the placement and position of the patch
* To assess preliminary efficacy based on:
* Evaluation of visual function
* Eye fundus
* Evaluation of photoreceptor survival

Assessment of visual function by Diagnosys-Full-field stimulus threshold (D-FST) is the only exploratory objective.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of retinitis pigmentosa based on a genetic test confirming the presence of a monogenic mutation that affects a gene involved in the visual signalling process specifically at the level of RPEs, namely RPE65 or LRAT, or MerTK
* 18 years old ≤ Age ≤ 65 years old

For patient of the first cohort:

* Visual acuity ≤ 20/200 in the best eye (legally blind)

  - For patient of the second cohort:
* 20/63 > Visual acuity > 20/200 in the worst eye And
* Visible photoreceptor outer nuclear layer (ONL) on a spectral domain optical coherence tomography (OCT) scan

For the two cohorts:

* Negative serum pregnancy test in women of childbearing potential (a woman who is two years post-menopausal confirmed by a physician or surgically sterile is not considered to be of childbearing potential)
* Female patients of childbearing potential (if sexually active), committed to use two methods of contraception starting from the enrollment, during Mycophenolate Mofetil (MMF) treatment and for 6 weeks after the last dose of MMF
* Sexually active men (including vasectomized men) committed to use condoms during from the first day of MMF treatment and for at least 90 days after cessation of treatment
* Signed informed consents by the patient or legal guardian(s). For patients unable to give consent, authorization to participate to the study will be collected close to their legally authorized representative
* Affiliated to or a beneficiary of a health care system

Exclusion Criteria:

* - Patient unable or unwilling to comply with the protocol requirements
* History of allergy or sensitivity to one of the products used during the study
* Patients with known serious allergies to the fluorescein
* Patients with a contraindication to general anesthesia
* Prior treatment with a gene or cell therapy product
* Patients with chronic hepatitis B or C, i.e. positive hepatitis B surface antigen or hepatitis C RNA viral load positive
* Patients infected with Human immunodeficiency virus (HIV)
* Anti-HLA antibodies positive at screening
* Pregnancy or breastfeeding
* Presence of any ocular disease or ocular media opacity which in the opinion of the investigator precludes accurate evaluation
* Participation in another drug or device clinical study within last 6 months prior to baseline
* Patients known to be affected by pathologies for which the symptoms or associated treatments can alter the visual function and/or affect the retina
* Systemic corticosteroid therapy or other immunosuppressive / immunomodulating or anti-retroviral drugs within 2 months prior to baseline
* Patients with a contraindication to immunosuppressive/immunomodulating therapy (MMF) such as severe chronic renal impairment, severe digestive system disease, Lesch-Nyhan disease, Kelley-Seegmiller syndrome…
* Acute illness or infection within 4 weeks of the anticipated administration of study medication which may interfere with study assessments and immunosuppressive/immunomodulating therapy
* Any other condition or history that, in the opinion of the Investigator, may compromise the safety or compliance of the patient or would preclude the patient from successful completion of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Safety assessment | From Baseline until Week 56
  Safety and tolerability measured by the incidence of Adverse Events or Serious Adverse Events throughout the study

SECONDARY OUTCOMES:
Position of therapeutic patch | From baseline until Week 56
  Position of the therapeutic patch by serial images assessment
Placement of the therapeutic patch | From Baseline until Week 56
  Placement of the therapeutic patch by serial spectral domain Ocular Coherence Tomography (OCT) scan at baseline and by study visit
Change in leakage or perfusion | At baseline and weeks 24, 48, and 56
  Change in leakage or perfusion in normal fundal vasculature and presence of abnormal vasculature by fundus fluorescein angiography
Change in thickness of RPE layer | At weeks 4, 8, 16, 24, 36, 48 and 56
  Change in thickness of RPE layer by B-mode orbital ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane BERTIN, MD, Principal Investigator — Centre des 15-20
Locations (1):
- •Centre Hospitalier National d'Ophtalmologie (CHNO) des Quinze-Vingts, Paris, France

IPD SHARING:
Plan to Share IPD: No